CLINICAL TRIAL: NCT03790306
Title: Opioid Free and Therapy Minimized Advantages Using HANA Table for Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: St. Elizabeth Medical Center, Utica, NY (Other)
Responsible Party: Principal Investigator, Dr Andrew B. Wickline, Orthopedic Surgeon, St. Elizabeth Medical Center, Utica, NY
Other Study IDs: QIIIS
Record Dates: First submitted 2018-12-20; First posted 2018-12-31 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Arthropathy of Hip Joint; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To prove that anterior approach total hip arthroplasty using the HANA table can be performed with little, if any, need for opioids using a combination of education, optimized pre op and post op pain protocols and optimized recovery tools.

DETAILED DESCRIPTION:
Methods:

Data Collection:

* pre-op assessment/physical therapy evaluation
* post op assessment - PACU, phase II (Prior to discharge)
* phone calls after discharge (post op day 1, 2, 3)
* follow up assessment in surgeon's office (3 and 6 weeks post op)
* Ortech
* Swiftpath
* HOOS jr

Pre-optimization:

* All patients enroll in SwiftPath education program
* Optimized BMI, hemoglobin, albumin, glucose control, A1C and blood pressure control

Total Joint procedure:

-anterior approach using the HANA table THA preformed with intra-articular block

Pain Management regimen:

* Pre op PT teaching
* post op multimodal pain regimen

ELIGIBILITY:
Inclusion Criteria:

* Elective total hip arthroplasty
* unilateral
* patient surgeries scheduled to be performed at the hospital and surgery center
* patients must enroll in SwiftPath
* Ability to read and understand English

Exclusion Criteria:

* Patient diagnosis of schizophrenia, bipolar disease, dementia
* previous burn to affected extremity
* BMI > 40
* Hemoglobin <12 female, <13 male
* Albumin less than 3.5
* A1C >8.0

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females presenting seeking elective unilateral total hip arthoplasty that fall within inclusion criteria listed above
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wickline, MD, Principal Investigator — St. Elizabeth's Medical Center
Locations (1):
- St. Elizabeth's Medical Center, Utica, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- THR With HANA Table: Patients undergoing Total Hip Replacement (THR) with use of the Hip And kNee Arthroplasty (HANA) table.
Period: Overall Study
Arm/Group | THR With HANA Table
Started | 207
Completed | 207
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 202
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 207

OUTCOME MEASURES:

1. Primary Outcome: Pre-operative Narcotic Use
Description: Percentage of patients that used used opioids pre-operatively
Time Frame: Pre-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
Participants | 30

2. Primary Outcome: Number of Patients That Took Any Opioids Throughout 6-week Follow-up Period
Description: Number of patients that took any opioids throughout 6-week follow-up period
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
Participants | 128

3. Primary Outcome: Short Physical Performance Battery
Description: Assessment tool measuring gait speed, balance and chair stand test. Scores range from 0 to 4 with higher scores indicating a better outcome.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
score on a scale
  Balance | 3.95 (0.31)
  Gait | 3.89 (0.45)
  Chair | 3.17 (1.31)

4. Secondary Outcome: Numeric Pain Scores
Description: A numeric pain score (0-10, 0 is no pain and 10 is worst imaginable pain). This will be used to assess patients level of pain relating to opioid use and recovery. Both 'best' pain level and 'worst' pain level as reported by the patient will be reported.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
units on a scale
  Best pain level | 0.00966 (0.139)
  Worst pain level | 2.14 (1.77)

5. Secondary Outcome: Sleep Quality
Description: The percentage of patients where pain interrupts sleep 'never' or 'rarely' will be combined together and reported.
Time Frame: 6 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
Participants | 184

6. Secondary Outcome: Number of Participants Who Adhere to Prescribed Post op Recovery Protocol
Description: Number of Participants Who Adhere to Prescribed Post op Recovery Protocol collected via a questionnaire
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
Participants | 206

7. Secondary Outcome: Length of Stay in Hospital
Description: Average number of days in hospital after surgery
Time Frame: 1 week
Measure: Mean (Full Range); unit: days
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
days | 0.4175 [0 to 6]

8. Secondary Outcome: Number of Patients That Return to Work 6 Weeks After Surgery
Description: questionnaire asking the patient to report whether or not they have returned to employment and at what capacity (using Department of Labor physical employment scale). Patients will answer "yes" or "no" when asked if they have returned to work.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- THR With HANA Table: Patients undergoing Total Hip Replacement (THR) using the Hip And kNee Arthroplasty (HANA) table
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
Participants | 56

9. Secondary Outcome: Number of Patients Who Return to Driving 6 Weeks After Surgery
Description: Patients will respond yes or no when asked if they have resumed driving.
Time Frame: 6 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | THR With HANA Table
Number analyzed (Participants) | 207
Participants | 182

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | THR With HANA Table
All-Cause Mortality (participants affected / at risk) | 0/207
Serious Adverse Events (participants affected / at risk) | 0/207
Other Adverse Events (participants affected / at risk) | 0/207

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03790306/Prot_SAP_000.pdf